## Consent Form - Clinic Personnel

COMIRB APPROVED For Use 29-Nov-2022 15-Jun-2023

Principal Investigator: Monica Perez Jolles, PhD

COMIRB No: 22-0547 Version Date: 11/29/2022

**Study Title:** Supporting the implementation of a state policy on screening for

Adverse Childhood Experiences (ACEs) in Federally Qualified Health

Centers.

You are being asked to be in a research study. This form provides you with information about the study. A member of the research team will describe this study to you and answer all of your questions. Please read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

# Why is this study being done?

The purpose of this study is to support Borrego Health in the implementation of the Adverse Childhood Experiences or ACEs Aware state program screening children for adverse childhood experiences. You are being asked to take part in this study because you are a staff member /provider/manager at one of the Borrego Health clinics and are involved in some way with the implementation of the California ACEs Aware screening program. Up to 80-100 clinic staff will participate in the study.

## What happens if I join this study?

If you join the study, you will receive a link to a short survey online. Questions will be related to your views on challenges and facilitators to implementing the ACEs screenings in clinical settings. A basic demographic questionnaire will be included at the end. No names will be included in the survey. This should take about 10-15 minutes. We will randomly select six survey participants from each participating clinic to participate in a follow-up interview. If selected and within days of receiving the link, you will also be contacted by the research team to invite you to participate in a 30-45 minute phone interview. Questions will relate to your views on the feasibility of the ACEs screenings, your satisfaction with the support provided by Borrego Health's implementation coach, and a trauma-informed workgroup.

## What are the possible discomforts or risks?

Discomforts you may experience while in this study include that a question may make you feel uneasy or embarrassed. You can choose to skip or stop answering any questions you don't want to. Other possible risks include a small risk that people who are not connected with this study will learn your identity or your personal information.

#### What are the possible benefits of the study?

There are no direct benefits to you from taking part in this study. This study is designed for the researcher to learn more about how clinics can best implement ACEs screenings for children

### Consent Form - Clinic Personnel

and for the benefit of other pediatric patients. There are also benefits to communities and society as gained knowledge.

# Who is paying for this study?

This research is being paid for by the National Institute of Mental Health.

# Will I be paid for being in the study? Will I have to pay for anything?

You will be paid a \$25 gift card the first time you take the survey, and an additional \$25 gift card if you are invited to participate in the follow-up interview.

### Is my participation voluntary?

Taking part in this study is voluntary. You have the right to choose not to take part in this study. If you choose to take part, you have the right to stop at any time. If you refuse or decide to withdraw later, you will not lose any benefits or rights to which you are entitled.

# Who do I call if I have questions?

The researcher carrying out this study is Monica Perez Jolles, Ph.D. You may ask any questions you have now. If you have questions later, you may call Monica Perez Jolles at 303.724.0829. You may have questions about your rights as someone in this study. You can call Monica Perez Jolles with questions. You can also call the Multiple Institutional Review Board (IRB). You can call them at 303-724-1055.

#### **Certificate of Confidentiality**

This study has been issued a Certificate of Confidentiality from the federal government to help protect your privacy. The Certificate prohibits the researchers from disclosing your name, or any identifiable information, document or biospecimen from the research, with the exceptions listed below. A certificate provides protections against disclosing research information in federal, state, or local civil, criminal, administrative, legislative or other proceedings.

These protections apply only to your research records. The protections do not apply to your medical records.

The researchers may disclose your name or identifiable information, document or biospecimen, under the following circumstances:

To those connected with the research,

If required by Federal, State or local laws,

If necessary for your medical treatment, with your consent,

For other scientific research conducted in compliance with Federal regulations,

To comply with mandated reporting, such as a possible threat to harm yourself or others, reports of child abuse, and required communicable disease reporting, or

Under other circumstances with your consent.

A Certificate of Confidentiality does not protect the information you or a member of your family voluntarily release.

#### Who will see my research information?

We will do everything we can to keep your records a secret. It cannot be guaranteed.

### Consent Form - Clinic Personnel

Both the records that identify you and the consent form signed by you may be looked at by others.

Federal agencies that monitor human subject research

Human Subject Research Committee

The group doing the study

The group paying for the study

Regulatory officials from the institution where the research is being conducted who want to make sure the research is safe

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

The results from the research may be shared at a meeting. The results from the research may be in published articles. Your name will be kept private when information is presented.

Recordings of interviews will be kept in a password-protected computer drive and they will be destroyed after the transcription has been finalized. All transcriptions will not include individual names or identifiable information. Transcriptions will be kept for 3 years, and then erased.

## Agreement to be in this study

I have read this paper about the study or it was read to me. I understand the possible risks and benefits of this study. I know that being in this study is voluntary. I choose to be in this study: I will get a copy of this consent form.

| Signature: | Date: |
|----------------------------|-------|
| Print Name: | |
| Consent form explained by: | Date: |
| Print Name | |